CLINICAL TRIAL: NCT04236661
Title: Reports on Sleep Quality and Thermoregulation Among Veterans
Acronym: ReSQuTheVets
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study team unable to start up study at this time
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: New Chilipad
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2019-12

CONDITIONS: Sleep Disturbance
Keywords: chilipad; Sleep disorders
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Twenty subjects with self-reporting sleep disturbance will use the Chilipad cooling mattress for 5 weeks. The subjects will be given a Diary to complete tracking sleep quality during the 5 weeks. Subjects will also be given questionnaires before and after the sleep study part of the study to measure changes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Chilipad Arm (Experimental): Subjects will use chilipad nightly for 5 weeks
  Interventions: Device: chilipad

INTERVENTIONS:
Device: chilipad — Chilipad is a commercially available pad designed to be placed between the top of a mattress and bed sheets. It allows for precise temperature regulation in one's bed.

SUMMARY:
To assess and compare the quality of sleep self- reported by veterans with sleep disorders before and after use of the Chilipad cooling mattress pad

DETAILED DESCRIPTION:
A non-randomized convenience sampling study of N=20 adult male or female veterans (> 18 years of age) with self-reporting sleep disturbance and will utilize a Chilipad cooling mattress for the 5-week study period

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female veteran patients (> 18 years of age)
* Self-report of sleep disturbance, defined as "sleep of poor quality, timing, efficiency, or duration"

Exclusion Criteria:

* Non-adult patients < 18 years of age.
* Patients with chart documentation or self-report of illegal drug use, impaired orientation and cognition or currently incarcerated.
* Initiated CAM or non-CAM treatments for sleep disturbance in the last 4 weeks.
* Changed dose of a CAM or non-CAM treatments for sleep disturbance in the last 4 weeks.
* Initiated antidepressants in the last 3 months.
* Changed of an antidepressant in the last 3 months.
* Patients who describe their health as fair or poor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep Related Impairment Short Form | 5-week prior intervention
  PROMIS sleep related impairment short form is a questionnaire with 8-item 5-point Likert rating scale survey reflecting DSM-5 for sleep disturbance. The raw score on 8 items is determined, summed for a raw score, then a T-score table is utilized to compare with the subject's individual score. The result, rounded to the nearest whole number determines the score. The survey T-scores are interpreted as: < 55 = none to slight; 55.0 - 59.9 = mild; 60.0 - 69.9 = moderate; and > 70 = severe
PROMIS Sleep Related Impairment Short Form | 5-week after intervention
  PROMIS sleep related impairment short form is a questionnaire with 8-item 5-point Likert rating scale survey reflecting DSM-5 for sleep disturbance. The raw score on 8 items is determined, summed for a raw score, then a T-score table is utilized to compare with the subject's individual score. The result, rounded to the nearest whole number determines the score. The survey T-scores are interpreted as: < 55 = none to slight; 55.0 - 59.9 = mild; 60.0 - 69.9 = moderate; and > 70 = severe

SECONDARY OUTCOMES:
OURA ring total sleep metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The total sleep metric will show hours of sleep each night.
OURA ring REM metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The total REM metric will show the total amount of REM sleep each night.
OURA ring DEEP sleep metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The DEEP sleep metric will show the number of hours of deep sleep each night.
OURA ring Efficiency metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. Efficiency means the percentage of time spent sleeping while in bed.
OURA ring latency metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. Latency is the amount of time it takes a study participant to fall to sleep.
OURA ring timing metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The timing records individual circadian rhythms.
OURA ring sleep score metric | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The sleep score metric will be determined by total sleep, efficiency, disturbances, REM sleep, deep sleep, sleep latency, sleep timing and light sleep.The sleep score ranges from 0-100. Higher scores denotes better outcomes.
OURA ring resting heart rate | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The resting heart rate will be recorded.
OURA ring respiration rate | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The respiration rate will be recorded.
OURA ring readiness score | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The readiness score is calculated taking in account sleep balance, previous day activity, activity balance, body temperature, resting heart rate (rhr), recovery index . Score will be between 0 and 100. A lower score indicates a worse outcome.
OURA ring Skin temperature | Nightly for 5 weeks
  OURA is a ring that is worn on a finger and collects information about the quality and duration of sleep. The OURA ring will measure skin temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Remy Coeytaux, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: describes oura ring outcome measures in detail — https://ouraring.com/